CLINICAL TRIAL: NCT07219810
Title: Accelerated iTBS Targeting of Working Memory Versus Inhibitory Control in Adolescent ADHD
Acronym: WINK
Status: Recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Bradley Hospital (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 2323018
Record Dates: First submitted 2025-09-03; First posted 2025-10-22 (Actual); Last update posted 2025-10-22 (Actual); Status verified 2025-09

CONDITIONS: ADHD
MeSH Terms: conditions — Attention Deficit Disorder with Hyperactivity

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- iTBS to the left DLPFC (Experimental)
  Interventions: Device: intermittent theta burst stimulation (iTBS)
- iTBS to the right pre-SMA (Active Comparator)
  Interventions: Device: intermittent theta burst stimulation (iTBS)

INTERVENTIONS:
Device: intermittent theta burst stimulation (iTBS) — Device: Stimulation will be delivered using a Nexstim NBT System 2 device. Motor Threshold: The iTBS pulse intensity will be set at 80% of resting motor threshold (MT). The iTBS protocol will administer 2-second trains with an 8-second inter-burst interval for 1800 pulses [600 bursts]), in 50 Hz bursts at 5 Hz (i.e., 200 ms intervals). Each session will last approximately nine minutes. As three sessions will be administered per day, there will be a 20-30 minutes break between each of the nine-minute iTBS sessions. Magnetic pulses will be delivered in an MRI neuro-navigated manner using a cooled figure-eight coil. The PreSMA target will be approximately defined based on MNI coordinates: 13, 18, 62. The left DLPFC target will be approximately defined based on MNI coordinates: -44, 28, 16.

SUMMARY:
The objective of this project is to examine the differential therapeutic effect of intermittent theta burst stimulation (iTBS; a type of repetitive transcranial magnetic stimulation) to the left DLPFC versus right PreSMA in modulating working memory (WM) versus inhibitory control (IC) deficits. Fifty adolescents (12-18 years old) with parent-reported WM and IC deficits and diagnosed ADHD will be randomized to DLPFC or PreSMA targeted 3x-daily iTBS for a total of ten days (30 total sessions).

ELIGIBILITY:
Inclusion Criteria

1. Age 12-18 years
2. English fluency of participant and parent and able to provide informed consent/assent
3. Clinical diagnosis of ADHD and confirmation of diagnostic criteria on the Diagnostic Interview for Anxiety, Mood, and OCD and Related Neuropsychiatric Disorders, Child and Adolescent Version (DIAMOND-KID)
4. Parent rating on The Behavior Rating Inventory of Executive Function-Second Edition (BRIEF-2), Parent Form: Working Memory scale T-Score > 60 AND Inhibition scale T-Score > 60
5. IQ > 70

Exclusion Criteria

Participants will be screened to exclude individuals with neurological or medical conditions that might confound the results, as well as to exclude participants in whom MRI or TMS might result in increased risk of side effects or complications. Common contraindications include metallic hardware in the body, cardiac pacemaker, patients with an implanted medication pumps or an intracardiac line, or prescription of medications known to lower seizure threshold. These account for most of the exclusion criteria listed below:

1. Intracranial pathology from a known genetic disorder (e.g., NF1, tuberous sclerosis) or from acquired neurologic disease (e.g. stroke, tumor), cerebral palsy, history of severe head injury, or significant dysmorphology
2. History of fainting spells of unknown or undetermined etiology that might constitute seizures
3. History of seizures, diagnosis of epilepsy, or immediate (1st degree relative) family history epilepsy
4. Any progressive (e.g., neurodegenerative) neurological disorder
5. Chronic (particularly) uncontrolled medical conditions that may cause a medical emergency in case of a provoked seizure (cardiac malformation, cardiac dysrhythmia, asthma, etc.)
6. Contraindicated metal implants in the head, brain or spinal cord (excluding dental implants or fillings)
7. Non-removable makeup or piercings
8. Pacemaker, implanted medication pump, or ventriculo-peritoneal shunt
9. Vagal nerve stimulator, deep brain stimulator, or transcutaneous electrical nerve stimulation unit
10. Signs of increased intracranial pressure
11. Intracranial lesion
12. History of head injury resulting in prolonged loss of consciousness
13. Substance abuse or dependence within past six months (i.e., DSM-5 substance use disorder criteria)
14. Chronic treatment with prescription medications that decrease cortical seizure threshold, not including psychostimulant medication if deemed to be medically safe as part of the medical review process.
15. Active psychosis or mania
16. Acute suicidal intent
17. Current pregnancy
18. Significant visual, hearing or speech impairment
19. Dental braces
20. Current wards of the state

Ages: 12 Years to 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 50 (Estimated)
Dates: Start 2025-09-01 (Actual); Primary Completion 2029-09-01 (Estimated); Study Completion 2029-09-01 (Estimated)

PRIMARY OUTCOMES:
EEG, source-localized oscillatory beta band bursting during SST/SWMT | Visit 13, approximately 1-2 days after iTBS
  PreSMA-targeted iTBS will lead to greater relative activation of the IC network versus the WM network (and the opposite pattern for DLPFC-targeted iTBS).
fMRI-measured blood oxygenation level-dependent (BOLD) activity during SST/NBT | Visit 13, approximately 1-2 days after iTBS
  PreSMA-targeted iTBS will lead to greater relative activation of the IC network versus the WM network (and the opposite pattern for DLPFC-targeted iTBS).
Task-based WM/IC performance on SWMT/N-Back/SST | Visit 13, approximately 1-2 days after iTBS
  PreSMA-targeted iTBS will lead to greater relative improvement of IC versus WM (and the opposite pattern for DLPFC-targeted iTBS)
Rater-Based WM/IC symptoms (BRIEF-2) | Visit 13, approximately 1-2 days after iTBS
  PreSMA-targeted iTBS will lead to greater relative improvement of IC versus WM (and the opposite pattern for DLPFC-targeted iTBS)

CONTACTS AND LOCATIONS:
Locations (1):
- E. P. Bradley Hospital, East Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Undecided